CLINICAL TRIAL: NCT02074709
Title: Transversus Abdominis Plane (TAP) Block With Bupivacaine Versus Wound Infiltration With Liposomal Bupivacaine (Exparel) for Postoperative Pain Management After Open Total Abdominal Hysterectomy: a Prospective Randomized Controlled Trial
Brief Title: TAP Block With Plain Bupivacaine Versus Wound Infiltration With Exparel for Postoperative Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Irina Gasanova, MD, PhD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 072013-080
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Pain
Keywords: Pain, Liposomal bupivacaine, Wound infiltration
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP block (Active Comparator): TAP block with plain bupivacaine
  Interventions: Drug: Plain bupivacaine
- Wound infiltration (Active Comparator): Wound infiltration with liposomal bupivacaine
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Plain bupivacaine — Intraoperative: TAP block with plain bupivacaine + Acetaminophen 1000 mg IV + Ketorolac 30 mg IV .
  First 24-h Postoperative: Ketorolac 30 mg, IV 3 more doses, + acetaminophen 1000 mg 3 more doses, + IV-PCA morphine.
  24-48-h Postoperative: Oral ibuprofen 800 mg q 8 h + hydrocodone/acetaminophen 5mg/500 mg 1-2 tablets q 6h,prn
  Other Names: Bupivacaine Hydrochloride
  Arms: TAP block
Drug: Liposomal bupivacaine — Group intraoperative: Wound infiltration with liposomal bupivacaine (Exparel) + IV acetaminophen 1000 mg IV + Ketorolac 30 mg IV
  First 24-h Postoperative: Ketorolac 30 mg, IV 3 more doses, + acetaminophen 1000 mg 3 more doses, + IV-PCA morphine
  24-48-h Postoperative: Oral ibuprofen 800 mg q 8 h + hydrocodone/acetaminophen 5mg/500 mg 1-2 tablets q 6h, prn
  Other Names: Exparel
  Arms: Wound infiltration

SUMMARY:
In this randomized, controlled, observer-blinded study we plan to evaluate pain relief after ultrasound-guided transversus abdominis plane (TAP) block using bupivacaine and wound infiltration using liposomal bupivacaine in patients undergoing abdominal hysterectomy.

DETAILED DESCRIPTION:
Patients undergoing open total abdominal hysterectomy at Parkland Hospital (n=60) will be randomized into one of two groups to receive either ultrasound-guided bilateral TAP block with bupivacaine (Group 1) or infiltration of the surgical wound with liposomal bupivacaine (Group 2) for postoperative pain management. The remaining aspect of perioperative care, including the general anesthetic technique, postoperative care will be standardized and will be similar for all patients. The duration of the involvement in the study will be until 48 hours postoperatively. The pre-anesthesia care unit personnel will identify patients during their preoperative clinic visit.

Patients in Group 1 will receive ultrasound-guided bilateral TAP block at the end of the surgery. Patients in Group 2 will receive Exparel prior to closing the incision which will be injected subfascially and subcutaneously. In the first 24-h postoperative period, patients in both Groups will receive acetaminophen 1000 mg every 6 h orally, ketorolac 30 mg, IV every 6 h, orally and morphine via an intravenous patient controlled analgesia (IV-PCA) system to maintain adequate pain control. In the 24-48 h study period, all patients will receive oral ibuprofen 800 mg and acetaminophen 1000 mg three times a day and a combination of hydrocodone/acetaminophen 5mg/ 325 mg 1-2 tablets, as needed.

The postoperative analgesia will be documented using the visual analog score (0=no pain, 10=worst pain). In addition, total opioid dose over the 48-h study period will be documented. Postoperative nausea will be measured using a categorical scoring system (none=0, mild=1, moderate=2, severe=3) and episodes of vomiting will be documented. Rescue antiemetics will be given to any patient who complains of nausea and/or vomiting.

All variables will be assessed at 2, 6, 12, 24, and 48 hours, postoperatively by an investigator blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Female
* ASA physical status 1-3
* Scheduled for open abdominal hysterectomy
* Age 18-80 years old
* Able to participate personally or by legal representative in informed consent in English or Spanish

Exclusion Criteria:

* History of relevant drug allergy
* Age less than 18 or greater than 80 years
* Chronic opioid use or drug abuse
* Significant psychiatric disturbance
* Inability to understand the study protocol
* Refusal to provide written consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irina Gasanova, MD., PhD., Principal Investigator — UTexas Southwestern Medical Center
Locations (1):
- UTSW, Parkland Health Hospital System, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 67 patients were assessed for eligibility and 60 patient enrolled to the study.
Groups:
- TAP Block: TAP block with plain bupivacaine
  Plain bupivacaine: Intraoperative: TAP block with plain bupivacaine + Acetaminophen 1000 mg IV + Ketorolac 30 mg IV .
  First 24-h Postoperative: Ketorolac 30 mg, IV 3 more doses, + acetaminophen 1000 mg 3 more doses, + IV-PCA morphine.
  24-48-h Postoperative: Oral ibuprofen 800 mg q 8 h + hydrocodone/acetaminophen 5mg/500 mg 1-2 tablets q 6h,prn
- Wound Infiltration: Wound infiltration with liposomal bupivacaine
  Liposomal bupivacaine: Group intraoperative: Wound infiltration with liposomal bupivacaine (Exparel) + IV acetaminophen 1000 mg IV + Ketorolac 30 mg IV
  First 24-h Postoperative: Ketorolac 30 mg, IV 3 more doses, + acetaminophen 1000 mg 3 more doses, + IV-PCA morphine
  24-48-h Postoperative: Oral ibuprofen 800 mg q 8 h + hydrocodone/acetaminophen 5mg/500 mg 1-2 tablets q 6h, prn
Period: Overall Study
Arm/Group | TAP Block | Wound Infiltration
Started | 30 | 30
Completed | 29 | 29
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Patient undergoing hysterectomy
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP Block | Wound Infiltration | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (6.4) | 44.4 (6.1) | 44 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Score on Coughing at 6 hr
Description: Visual Analog Pain Scores (VAS); 0 (no pain) to 10 (worst possible pain)
Time Frame: Participants' pain score was assessed at 6 hr after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- TAP Block: TAP block with plain bupivacaine
  Plain bupivacaine: Intraoperative: TAP block with plain bupivacaine + Acetaminophen 1000 mg IV + Ketorolac 30 mg IV .
- Wound Infiltration: Wound infiltration with liposomal bupivacaine
  Liposomal bupivacaine: Group intraoperative: Wound infiltration with liposomal bupivacaine (Exparel) + IV acetaminophen 1000 mg IV + Ketorolac 30 mg IV
Arm/Group | TAP Block | Wound Infiltration
Number analyzed (Participants) | 29 | 29
units on a scale | 5.28 (2.45) | 3.59 (1.70)

ADVERSE EVENTS:
Arm/Group | TAP Block | Wound Infiltration
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes